CLINICAL TRIAL: NCT07168720
Title: Study on Pharmacokinetics and Clinical Efficacy of Dexmedetomidine Hydrochloride Microneedles(DEX) for Preoperative Sedation in Children
Brief Title: The Study is Being Conducted to Evaluate the Efficacy and Safety of Dexmedetomidine Hydrochloride Microneedles for Preoperative Sedation in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Novaken Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BOJI2025016LH
Record Dates: First submitted 2025-08-27; First posted 2025-09-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Preoperative Sedation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): 16 Participants will receive the Dexmedetomidine hydrochloride Microneedles identified in Part 1 of the study. Randomized in a 1:1 ratio through the randomization system, and assigned to medium-pressure group or low-pressure group. A total of 16 children with a high body weight (weight ≥ 19.4 kg) will be included. They will be randomly divided into a medium-pressure group and a low-pressure at a ratio of 1:1.
  Interventions: Drug: Dexmedetomidine hydrochloride Microneedles
- part2 (Experimental): Participants will receive the dose identified in Part 1 of the study. A total of 24 children with high body weight (weighing less than 19.4 kg) will be included. They will be randomly divided into the low dose group , the high dose group and placebo group at a ratio of 1:1:1. They will be given Dexmedetomidine hydrochloride Microneedles or placebo.
  Interventions: Drug: Dexmedetomidine hydrochloride Microneedles; Drug: placebo
- part3 (Experimental): Participants will receive the dose identified in Part 2 of the study. A total of 24 children with low body weight (weighing less than 19.4 kg) will be included. They will be randomly divided into the low dose group , the high dose group and placebo group at a ratio of 1:1:1. They will be given Dexmedetomidine hydrochloride Microneedles or placebo.
  Interventions: Drug: Dexmedetomidine hydrochloride Microneedles; Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine hydrochloride Microneedles — Randomized in a 1:1 ratio through the randomization system, and assigned to medium-pressure group or low-pressure group.
  Arms: Part 1
Drug: Dexmedetomidine hydrochloride Microneedles — In the high weight group, 8 subjects will receive a high dose of Dexmedetomidine hydrochloride Microneedles.
  In the high weight group, 8 subjects will receive a low dose of Dexmedetomidine hydrochloride Microneedles.
  Arms: part2
Drug: placebo — In the high weight group, 8 subjects will receive Dexmedetomidine hydrochloride Microneedles blank preparation.
  Arms: part2
Drug: Dexmedetomidine hydrochloride Microneedles — In the low weight group, 8 subjects will receive a low dose of Dexmedetomidine hydrochloride Microneedles.
  In the low weight group, 8 subjects will receive a high dose of Dexmedetomidine hydrochloride Microneedles.
  Arms: part3
Drug: Placebo — In the low weight group, 8 subjects will receive Dexmedetomidine hydrochloride Microneedles blank preparation.
  Arms: part3

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and the population pharmacokinetic characteristics of Dexmedetomidine Hydrochloride Microneedles for preoperative sedation in children

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo-controlled Phase IIa clinical trial, using Dexmedetomidine Hydrochloride Microneedles as an investigational drug and the Dexmedetomidine Hydrochloride Microneedles blank preparation as a comparator. After going through the confirmation of inclusion/exclusion criteria with signed subjects, they will have a procedure either of the two arms. The subjects should follow designated physician's instructions accurately during the clinical trial period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 years to 6 years (inclusive ), any genders;
* Body weight meeting the criteria:
* Scheduled to undergo general anesthesia for surgery/procedure
* American Society of Anesthesiologists（ASA） I~II
* Provide written informed consent from the legal guardian

Exclusion Criteria:

* Allergy to any component of the Dexmedetomidine Hydrochloride Microneedle Patch, history of allergy to other sedative drugs, or known allergy to α2-adrenergic receptor-related products or excipients;
* Having received other sedative-hypnotic or analgesic drugs prior to randomization, where the time since last dose is less than 7 half-lives;
* History of bronchial asthma, chronic respiratory diseases, or other severe respiratory system diseases;
* History of neurological diseases such as ischemic encephalopathy encephalopathy, craniocerebral injury, etc., which in the investigator's judgment may affect the evaluation of the investigational product;
* History of thoracic, cardiac, or brain surgery;
* Presence of large areas of skin damage or skin conditions unsuitable for topical patch application on the inner aspects of both forearms or the outer aspects of both thighs;
* Abnormal liver/kidney function test values (ALT or AST >1.5 times the upper limit of normal [ULN], or bilirubin >1.5 × ULN, or serum creatinine >1.5 × ULN);
* Severe cardiovascular diseases (e.g., fulminant myocarditis, high-grade or third-degree atrioventricular block, sick sinus syndrome, severe arrhythmia, cardiomyopathy, severe pulmonary hypertension, pulmonary atresia, heart failure);
* Anemia requiring treatment, as judged by the investigator (hemoglobin <80 g/L);
* Use of highly selective α2 agonists or antagonists prior to randomization, where the time since last dose is less than 7 half-lives;
* Participation in another clinical trial (meaning having received an investigational drug or device) within 3 months prior to screening;
* Presence of severe psychiatric illness at screening leading to inability or unwillingness to cooperate;
* Other situations deemed by the investigator as unsuitable for inclusion.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event and Serious Adverse Event | Day2
  Incidence rate of Adverse Event and Serious Adverse Event

SECONDARY OUTCOMES:
Maximum blood concentration | 0 to 4 hour after administration
  Maximum blood concentration
Ramsay scale | 0 minute to 45 minutes after administration
  Sedation level using the Ramsay scale. Ramsay Satisfaction defined as a scale of 1,2, 3, 4,5,6; the minimum value is 1 , the maximum value is 6, higher scores mean a better outcome.
Sedation Success Rate | 0 minute to 45 minutes after administration
  Proportion of subjects who will accomplish to start the anesthetic indcution or medical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jinan University (Guangzhou Overseas Chinese Hospital), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: ICF
Time Frame: Data are available 6 months after the primary publication
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.novaken.cn/